CLINICAL TRIAL: NCT02296996
Title: A Phase II Clinical Trial on the Combination of Dabrafenib and Trametinib for BRAF-inhibitor Pretreated Patients With Advanced BRAF V600 Mutant Melanoma
Brief Title: Dabrafenib and Trametinib for BRAF-inhibitor Pretreated Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Bart Neyns, Bart Neyns, MD PhD, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UZB-BN- 2013-001
Record Dates: First submitted 2014-10-15; First posted 2014-11-21 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Malignant Melanoma
Keywords: BRAF V600; Rechallenge; Combination; Dabrafenib; Trametinib
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dabrafenib + trametinib (Experimental): Single arm study with dabrafenib + trametinib combination therapy
  Interventions: Drug: Dabrafenib + Trametinib

INTERVENTIONS:
Drug: Dabrafenib + Trametinib

SUMMARY:
Patients with BRAF V600 mutant advanced melanoma benefit from treatment with a BRAF-inhibitor (e.g. dabrafenib, vemurafenib) and from combination of a BRAF- and MEK-inhibitor (e.g. dabrafenib and trametinib). Following initial tumor regression, progression is diagnosed in a majority of patients treated with BRAF-inhibitor mono-therapy within the first 12-months of therapy. Various molecular mechanisms that underlie the development of resistance to treatment with a BRAF-inhibitor have been reported. These mechanisms do not include secondary mutations in the BRAF-gene and therefore resistance to BRAF-inhibition could potentially be reversible when selective pressure by BRAF-inhibition is withheld for a sufficient period of time of melanoma progression. This clinical trial protocol addresses the potential renewed anti-tumor activity of combined BRAF- and MEK inhibition with the combination of dabrafenib and trametinib in patients with unresectable AJCC stage III or - IV BRAF V600 mutant melanoma who are documented with progression of disease at least 12 weeks following the last day of dosing of a BRAFinhibitor containing treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and signed written informed consent.
2. Histologically confirmed cutaneous melanoma that is either Stage IIIC (unresectable) or Stage IV (metastatic), and determined to be BRAF V600E/K mutation-positive.
3. Subjects must have failed at least two prior systemic anti-cancer treatments for Stage IIIC (unresectable) or Stage IV (metastatic) melanoma that must have included:

   * Treatment with a BRAF inhibitor (including but not limited to dabrafenib, vemurafenib, and LGX818) and progression of disease per RECIST, version 1.1 [Eisenhauer, 2009] must have been documented during this treatment.
   * Treatment with ipilimumab (or an alternative experimental immunotherapy) and progression of disease per immune related response criteria [Wolchock Clin Cancer Res December 1, 2009 15; 7412] must have been documented during this treatment.
4. Documented progression of disease per RECIST, version 1.1 [Eisenhauer, 2009]) or per immune related response criteria [Wolchock Clin Cancer Res December 1, 2009 15; 7412] if the latest systemic therapy administered was ipilimumab, an anti-PD1 or anti-PD-L1 therapy, or any other experimental immunotherapy.
5. The presence of at least one measurable lesion per RECIST, version 1.1 [Eisenhauer, 2009]).
6. Interval between the date of the last administration of prior therapy for melanoma and the date of recruitment:

   * > 12 weeks following the date of the last administration of a BRAF-inhibitor;
   * > 12 weeks following the date of the first administration and > 4 weeks following the date of the last administration of ipilimumab, or an anti-PD1, or anti-PD-L1 therapy;
   * > 4 weeks following the date of the last administration of chemotherapy (> 6 weeks in case of a nitrosurea or mitomycin C containing regimen);
   * > 4 weeks following major surgery or extensive radiotherapy.
7. Subjects with ocular melanoma are not eligible.
8. All prior anti-cancer treatment-related toxicities (except alopecia and laboratory values as listed on Table 2) must be ≤ Grade 1 according to the Common Terminology Criteria for Adverse Events version 4 (CTCAE version 4.0; National Cancer Institute ( NCI,) 2009) at the time of recruitment.
9. Able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
10. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to recruitment and agree to use effective contraception, as defined in Section 7.3.3.1, throughout the treatment period, and for 4 months after the last dose of study treatment.
11. An Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 [Oken, 1982]. Refer to Appendix 1 for details.
12. Adequate baseline organ function as defined in Table 2.

Exclusion Criteria:

1. Grade 4 or repetitive grade 3 adverse event(s) related to prior treatment with a BRAF- and/or MEK inhibitor.
2. Any contra-indication for evaluation by whole body CT and MRI of the brain.
3. Taken an investigational drug within 28 days or 5 half-lives (minimum 14 days), whichever is shorter, prior to recruitment.
4. Current use of a prohibited medication as described in Section 6 or requires any of these medications during treatment.
5. History of another malignancy, including any malignancy with confirmed activating RAS mutation. Note: Prospective RAS testing is not required. However, if the results of previous RAS testing are known, they must be used in assessing eligibility. Exception: Subjects who have been disease-free for 3 years, (i.e. subjects with second malignancies that are indolent or definitively treated at least 3 years ago) not including malignancy with confirmed activating RAS mutation, or subjects with a history of completely resected non-melanoma skin cancer.
6. Any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that could interfere with the subject's safety, obtaining informed consent, or compliance with study procedures.
7. Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (subjects with laboratory evidence of cleared HBV and HCV infection will be permitted).
8. Patients with progressive symptoms from active brain metastasis or in need of an increase in corticosteroids dose to control symptoms within 4 weeks prior to recruitment are excluded
9. No enzyme inducing anticonvulsants for ≥ 4 weeks prior to recruitment
10. A history or evidence of cardiovascular risk including any of the following:

    * Current LVEF < LLN
    * A QT interval corrected for heart rate using the Bazett's formula (QTcB; Section 5.6.3.3) ≥480 msec;
    * A history or evidence of current clinically significant uncontrolled arrhythmias; Exception: Subjects with atrial fibrillation controlled for > 30 days prior to recruitment are eligible.
    * A history (within 6 months prior to recruitment) of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty or stenting;
    * A history or evidence of current ≥Class II congestive heart failure as defined by the New York Heart Association (NYHA) guidelines (Appendix 4);
    * Treatment refractory hypertension defined as a blood pressure of systolic >140 mmHg and/or diastolic > 90 mm Hg which cannot be controlled by antihypertensive therapy;
    * Patients with intra-cardiac defibrillators;
    * Abnormal cardiac valve morphology (≥grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study.
11. Uncorrectable electrolyte abnormalities (e.g. hypokalaemia, hypomagnesaemia, hypocalcaemia), long QT syndrome or taking medicinal products known to prolong the QT interval.
12. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide (DMSO).
13. Females who are pregnant or nursing.
14. Interstitial lung disease or pneumonitis
15. Patients with a prior history of central serous retinopathy or retinal vein occlusion are excluded. Patients with a preexisting major ocular pathology are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Participants will be monitored until progression, with an expected average of 6 months

SECONDARY OUTCOMES:
Progression-free survival | Participants will be monitored until progression, with an expected average of 6 months
Overall Survival | 2 years
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Participants will be monitored until progression, with an expected average of 6 months
  Detect adverse events

OTHER OUTCOMES:
Tumour-specific cfDNA levels | Participants will be monitored until progression, with an expected average of 6 months
  To explore if tumor specific cfDNA levels can be used as a monitoring tool to detect early progression of disease

CONTACTS AND LOCATIONS:
Overall Officials: Neyns Bart, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Brussels, Belgium

REFERENCES:
- [Derived] Schreuer M, Jansen Y, Planken S, Chevolet I, Seremet T, Kruse V, Neyns B. Combination of dabrafenib plus trametinib for BRAF and MEK inhibitor pretreated patients with advanced BRAFV600-mutant melanoma: an open-label, single arm, dual-centre, phase 2 clinical trial. Lancet Oncol. 2017 Apr;18(4):464-472. doi: 10.1016/S1470-2045(17)30171-7. Epub 2017 Mar 4. PMID 28268064